CLINICAL TRIAL: NCT03032796
Title: Characterizing the Synergistic Effects of Physical and Cognitive Training on Attention and Working Memory
Acronym: BBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1R21MH110743-01
Record Dates: First submitted 2017-01-12; First posted 2017-01-26 (Estimated); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Healthy Adults

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BBT (Experimental): Body-Brain Trainer
  Interventions: Behavioral: Body-Brain Trainer
- Body Trainer (Active Comparator): Participants will only perform a basic reaction task in each level/module to ensure only the most minimal cognitive challenge is present, while completing all of the physical aspects of BBT. Thus this will be a physical training protocol.
  Interventions: Behavioral: Body Trainer
- Brain Trainer (Active Comparator): The "Brain Trainer" group will train using the same platform as the BBT group, except while sitting down and playing with an Xbox control pad (thus removing all physical training aspects).
  Interventions: Behavioral: Brain Trainer
- Expectancy Matched Control Group (Placebo Comparator): The placebo-matched control group will engage in a battery of three apps in the laboratory that we believe will have no significant impact on cognition
  Interventions: Behavioral: Expectancy Matched Control

INTERVENTIONS:
Behavioral: Body-Brain Trainer — A novel video game-based intervention that incorporates i) adaptive algorithms critical for cognitive training, ii) physiological measures such as heart rate into the core game mechanics, and iii) motion capture technology to incorporate whole-body kinematics into game play. This group will train for 36 minutes per day, 3 days a week for 8 weeks.
  Arms: BBT
Behavioral: Body Trainer — A novel video game-based intervention that incorporates physiological measures such as heart rate into the core game mechanics, with motion capture technology to incorporate whole-body kinematics into game play. This group will train for 36 minutes per day, 3 days a week for 8 weeks. The "Body Trainer" group will train using closed-loop adaptive algorithms to challenge physical performance as guided by heart rate, such that the amount of movement needed to respond on each task will dynamically change depending upon the participant being below/above a predetermined derived level of exertion. During "Body Training", participants will only perform a basic reaction task in each level/module to ensure only the most minimal cognitive challenge is present
  Arms: Body Trainer
Behavioral: Brain Trainer — The "Brain Trainer" group will train using the aforementioned closed-loop adaptive algorithms to challenge cognitive performance, except while sitting down and playing with an Xbox control pad (thus removing all physical training aspects). This group will train for 36 minutes per day, 3 days a week for 8 weeks.
  Arms: Brain Trainer
Behavioral: Expectancy Matched Control — The placebo-matched control group will engage in a battery of three apps (playing each app 10 minutes per day, 5 days a week for 8 weeks completed in the laboratory that we believe will have no significant impact on the cognitive or physical fitness measures we are assessing: i) an app with 100 different logic games of varying difficulty and length, ii) a language-learning app with 10 language options, and iii) an app that offers a guided Tai Chi program. We have pre-determined that this approach generates matched expectancy compared to our training groups: we asked 100 naïve individuals to predict how they would expect to improve performance on our outcome measures after training on one of these platforms, revealing that placebo training generates equivalent expectations of improvement across each outcome measure as the BBT group.
  Arms: Expectancy Matched Control Group

SUMMARY:
The primary goal of this project is to evidence potential synergistic benefits on cognitive control processes using a video game ("Body-Brain Trainer", or BBT) that integrates cognitive and physical challenges in a complimentary fashion. Healthy adults will be recruited for a longitudinal experiment and randomly assigned to one of four study groups to mechanistically tease apart the possible presence of any synergistic effects on cognitive abilities through the combination of cognitive & physical challenges.

DETAILED DESCRIPTION:
Cognitive control functions (e.g. attention, working memory, goal-management) dictate our ability to learn and accomplish selected behavioral goals, with deficiencies in these processes found in a range of mental illnesses. The primary goal of this project is to evidence potential synergistic benefits on cognitive control processes using a video game ("Body-Brain Trainer", or BBT) that integrates cognitive and physical challenges in a complimentary fashion. Healthy adults will be recruited for a longitudinal experiment and randomly assigned to one of four study groups: 1) BBT, 2) "Brain Training" (BBT played with a gamepad controller), 3) "Body Training" (BBT without any cognitive demands), and 4) an expectancy matched placebo control group. Individuals will engage in eight weeks of training within our Neuroscape Laboratory, with pre- and post-training assessments evaluating physical, cognitive, and neural measures. The completion of this project will result in a more sophisticated understanding of how the integration of cognitive and physical training potentially impacts cognitive control processes, setting the stage for more effective interventions for mental illness and learning-related impairments.

ELIGIBILITY:
Inclusion Criteria:

* Can walk briskly for at least 15 minutes continuously without stopping
* Can stand up from a chair without using your hands
* Available to come 3x/week to our UCSF Mission Bay laboratory for 8 weeks
* Willing and able to undergo MRI, EEG procedures
* English fluency

Exclusion Criteria:

* cardiac problems
* bypass surgery
* pacemaker or heart valve replacement
* stroke
* respiratory conditions
* head trauma with loss of consciousness for less than a few minutes
* severe head trauma with loss of consciousness for more than a few minutes
* high/low blood pressure
* kidney failure
* electroconvulsive therapy (ECT)
* seizures
* implanted electrodes
* cancer/chemotherapy/radiation
* diabetes
* irritable bowel syndrome
* back problems
* claustrophobia
* Having been diagnosed with a psychiatric or neurological disorder
* Use of an assistive device (e.g., cane or walker) at any time to assist with ambulation
* Joint problems causing significant pain upon movement
* Heart Disease or Cardiovascular Disease
* Respiratory Disease (Lung Disease)

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-01; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin A. Anguera, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Neuroscape, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We were only able to enroll in 2 of the 4 arms for this study due to resource limitations for this study.
Groups:
- Body-Brain Trainer: Body-Brain Trainer
  Body-Brain Trainer: A novel video game-based intervention that incorporates i) adaptive algorithms critical for cognitive training, ii) physiological measures such as heart rate into the core game mechanics, and iii) motion capture technology to incorporate whole-body kinematics into game play. This group will train for 36 minutes per day, 3 days a week for 8 weeks.
Period: Overall Study
Arm/Group | Body-Brain Trainer | Expectancy Matched Control Group
Started | 24 | 25
Completed | 24 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Body-Brain Trainer | Expectancy Matched Control Group | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (5.9) | 68.2 (6.7) | 68.5 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 11 | 12 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 24 | 25 | 49
mCPT [Mean (Standard Deviation); unit: milliseconds] | 72.5 (39.7) | 52.2 (31.2) | 62.2 (35.5)
EEG [Mean (Standard Deviation); unit: decibles] | 0.77 (1.85) | 1.67 (2.27) | 1.33 (2.02)

OUTCOME MEASURES:

1. Primary Outcome: mCPT (Derived From Test of Variables of Attention (T.O.V.A.))
Description: A change from baseline regarding measurement of sustained attention and impulsivity abilities
Time Frame: At baseline and following the intervention (these data were collected no more than 1 week after intervention period ended, thus approximately 9 weeks after baseline data were collected)
Population: Due to logistical/practical consideration surrounding funding for this project, we were forced to only collect data for 2 gropus
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- BBT: Body-Brain Trainer: Body-Brain Trainer
  Body-Brain Trainer: A novel video game-based intervention that incorporates i) adaptive algorithms critical for cognitive training, ii) physiological measures such as heart rate into the core game mechanics, and iii) motion capture technology to incorporate whole-body kinematics into game play. This group will train for 36 minutes per day, 3 days a week for 8 weeks.
Arm/Group | BBT: Body-Brain Trainer | Body Trainer | Brain Trainer | Expectancy Matched Control Group
Number analyzed (Participants) | 24 | 0 | 0 | 25
milliseconds | 72.5 (39.7) |  |  | 52.2 (31.2)

2. Secondary Outcome: Delayed Recognition Working Memory Task: Response Time Variability Prior to and 9-weeks After Baseline
Description: A change from baseline regarding measurement of working memory abilities in the presence of interference. This task involved memorizing a face for set amount of time, followed by a delay period (during which participants were exposed to different types of distracting images), followed by the presentation of an image that participants are cued to respond whether or not this image matches the initial one presented. Here we examined a version of response time variance derived from exGaussain Statistics called tau, that is a measure of response time variance that considers the tails on a Gaussian distribution with respect to response time variability. This analysis allows one to see how variant one's performance could be on trials that fall outside of their mean performance distribution.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Body-Brain Trainer | Expectancy Matched Control Group
Number analyzed (Participants) | 24 | 25
msec | 29.7 (14.1) | 24.1 (10.0)

3. Other Pre Specified Outcome: Blood Pressure Measures
Description: Assessing a change in systolic & diastolic pressure following the intervention
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Body-Brain Trainer | Expectancy Matched Control Group
Number analyzed (Participants) | 24 | 25
mmHG | 78.72 (5.25) | 76.23 (5.91)

4. Other Pre Specified Outcome: Limit of Stability
Description: Assessing a change in balance following the intervention
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters/sec
Arm/Group | Body-Brain Trainer | Expectancy Matched Control Group
Number analyzed (Participants) | 24 | 25
meters/sec | 3.88 (1.34) | 4.29 (1.26)

5. Other Pre Specified Outcome: EEG Functional Measure (Event-related Spectral Perturbation)
Description: Assessing a change in event-related spectral perturbation following the intervention
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: dB (decibles)
Arm/Group | Body-Brain Trainer | Expectancy Matched Control Group
Number analyzed (Participants) | 24 | 25
dB (decibles) | .77 (1.85) | 1.67 (2.27)

6. Other Pre Specified Outcome: EEG Functional Measure (Long-range Coherence as Measured Via Phase Locking Values): Decibels Prior to and at 9 Weeks Post Baseline
Description: Assessing a change in coherence following the intervention. This measure assesses the synchronization of neural activity between frontal and posterior regions of the brain, looking to quantify how coherent these signals are. For example, if the activity at the front of the head shows greater synchrony with activity at the back of the head, than this measure of interest would show a greater amount of coherence.
  Coherence of this type is reported in the form of phase locking value, which tells us how consistently the timing of those rhythms stay aligned across many repetitions of the same event. PLV close to 1 (or 100%) → very consistent timing, almost perfectly locked together, whereas PLV close to 0 → timing is random, no consistent relationship. PLVs are typically reported in decibels to facilitate seeing subtle changes, compare across conditions, and stay consistent with other brainwave measures.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Decibels
Arm/Group | Body-Brain Trainer | Expectancy Matched Control Group
Number analyzed (Participants) | 24 | 25
Decibels | .24 (.09) | .28 (.09)

ADVERSE EVENTS:
Time Frame: Each participant was in the primary data collection period of the study for approximately 10 weeks (1 week for the collection of baseline measures, 8 weeks for training, and another week for the collection of post-training measures. There was a follow-up data collection 1 year following their post-training data collection to test for long-term beneficial effects. Thus the period of time over which we assessed for adverse events was 14.5 months in total.
Description: No difference in the definition of an adverse event from that listed at clinicaltrials.gov
Groups:
- BBT - Body-Brain Trainer: Body-Brain Trainer
  Body-Brain Trainer: A novel video game-based intervention that incorporates i) adaptive algorithms critical for cognitive training, ii) physiological measures such as heart rate into the core game mechanics, and iii) motion capture technology to incorporate whole-body kinematics into game play. This group will train for 36 minutes per day, 3 days a week for 8 weeks.
Arm/Group | BBT - Body-Brain Trainer | Body Trainer | Brain Trainer | Expectancy Matched Control Group
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/0 | 0/0 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/0 | 0/0 | 0/25
Other Adverse Events (participants affected / at risk) | 0/24 | 0/0 | 0/0 | 0/25

LIMITATIONS AND CAVEATS:
We were not able to collect all four arms as originally intended due to logistical and resource issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-06-18): https://cdn.clinicaltrials.gov/large-docs/96/NCT03032796/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/96/NCT03032796/SAP_001.pdf